CLINICAL TRIAL: NCT00162604
Title: Antibiotikaprofylakse Ved Vaginalplastik
Brief Title: Prophylactic Antibiotic Treatment During Vaginal Repair
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hvidovre University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2602-415
Record Dates: First submitted 2005-09-09; First posted 2005-09-13 (Estimated); Last update posted 2006-09-11 (Estimated); Status verified 2005-02

CONDITIONS: Uterine Prolapse; Cystocele; Rectocele; Enterocele
Keywords: Prophylactic antibiotic; Postoperative infections; Uterine prolapse grade I - II; cystocele; rectocele; enterocele; defects of the perineal body
MeSH Terms: conditions — Uterine Prolapse; Cystocele; Rectocele; Hernia | interventions — Cefuroxime

INTERVENTIONS:
Drug: Cefuroxime

SUMMARY:
Prolapse of the uterus, bladder and rectum is a common condition in multiparous and/or elderly women. The number of operations for vaginal repair is increasing in Denmark, but there is no consensus or evidence found about the efficiency of prophylactic antibiotics intraoperatively concerning postoperative infections.

The objective of this randomized, controlled trial is to investigate the significance of prophylactic antibiotic treatment in vaginal repair operations.

ELIGIBILITY:
Inclusion Criteria:

* Women ages 18+ with uterine prolapse grade I - II and/or cystocele and/or rectocele and/or enterocele grade I - II and/or defects of the perineal body, in whom there is medical indication for vaginal repair, but no indication for vaginal hysterectomy or transvaginal suspension of the vaginal vault after prior hysterectomy.

Exclusion Criteria:

* Patients allergic to cefuroxime.
* Patients in whom a vaginal hysterectomy or a transvaginal suspension of the vaginal vault or other major surgery is planned, where prophylactic antibiotic treatment is standard.
* Patients suffering from physical or mental disorders that will not allow them to give informed consent.
* Pregnant and nursing women.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 2005-05

PRIMARY OUTCOMES:
primary endpoint: no infections (urinary tract infections, pneumonia,wound infections, infected haematomas, etc.) within 30 days postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Marianne Ottesen, M.D, Ph.D, Study Director — Hvidovre University Hospital
Locations (1):
- Hvidovre University Hospital, Hvidovre, Denmark